CLINICAL TRIAL: NCT01689571
Title: A Randomised, Double-blind, Placebo-controlled, Three-way Crossover Study to Evaluate the Efficacy After Allergen Challenge, Safety and Tolerability of Two Doses of Inhaled CHF6001 DPI After 9 Days of Treatment in Adult Patients With Asthma
Brief Title: A Study to Evaluate the Efficacy After Allergen Challenge, Safety and Tolerability of Inhaled CHF6001 DPI in Asthmatics
Acronym: CHF6001_POC2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-1202-PR-0080; 2012-001483-29 (EudraCT Number)
Record Dates: First submitted 2012-09-04; First posted 2012-09-21 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: PDE4 inhibitor; Allergen Challenge; Asthma
MeSH Terms: conditions — Asthma | interventions — tanimilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo DPI (Placebo Comparator): Placebo by inhalation for 9 days
  Interventions: Drug: Placebo
- CHF6001 DPI Dose 2 (Experimental): CHF6001 by inhalation for 9 days
  Interventions: Drug: CHF6001
- CHF6001 DPI Dose1 (Experimental): CHF6001 by inhalation for 9 days
  Interventions: Drug: CHF6001

INTERVENTIONS:
Drug: CHF6001
  Arms: CHF6001 DPI Dose 2; CHF6001 DPI Dose1
Drug: Placebo
  Arms: Placebo DPI

SUMMARY:
The study is designed to look at the safety, tolerability and efficacy of 2 different doses of the study drug (CHF6001, a PDE4 inhibitor) in asthmatics, when given by inhalation, once a day for 9 days. The efficacy will be evaluated by measuring the protective effect of CHF 6001 after an allergen challenge.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent obtained
* Non smoking or ex-smokers from at least 1 year prior to study entry
* Males of females between 18 and 60 years inclusive
* Body Mass Index between 18 and 32 kg/m2
* Ability to be trained about the proper use of the inhalation device and to perform spirometry
* With mild to moderate allergic asthma as defined by the GINA guideline, steroid naive
* Atopy to at least one common aeroallergen
* Positive allergen-induced Early Asthmatic Response and Late Asthmatic Response at screening
* Ability to produce an adequate sputum sample
* Post-menopausal women, women of not childbearing potential or males and females of childbearing potential willing (they or their partner) to use a reliable method of contraception.

Exclusion Criteria:

* Worsening of asthma or respiratory tract infection prior to study entry
* History of life-threatening asthma or hospitalization for asthma prior to the study entry
* Pregnant or lactating women
* History of clinically significant hypotensive episodes or fainting, dizziness or light-headedness
* History or symptoms of clinically relevant neurologic disease
* Symptomatic hay fever
* Unstable concurrent disease that may impact the feasibility of the study
* Use of systemic corticosteroids, nebulised bronchodilator or oral beta2-agonist
* Use of leukotrienes modifiers, roflumilast or cromoglycate
* Use of long acting beta2-agonist or inhaled corticosteroids
* Use of short-acting or long-acting non-sedatives antihistamines
* Use of any other medication for the treatment of allergic asthma other than salbutamol
* Having received an investigational medicinal drug within 30 days prior to study entry
* Blood drawn of at least 250 ml in the previous 45 days
* Ongoing use of tobacco
* Other lung disease
* Recent history of alcohol dependency
* Inability to comply with the study protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Allergen challenge | after 9 days of treatment

SECONDARY OUTCOMES:
Induced Sputum | After 9 days of treatment
Methacholine challenge | After 9 days of treatment

OTHER OUTCOMES:
Pharmacokinetics of CHF6001 and its metabolites | after 9 days of treatment
  The following parameters will be evaluated at the steady state: AUC0-t, AUC0-24h, Cmax, Cmin, Cav, tmax, tmin, t½, CL/F and Vz/F
Vital signs | After single dose and 9 days of treatment
ECG | After single dose and 9 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Medicines Evaluation Unit; Brian Leaker, MD, Principal Investigator — Respiratory Clinical Trials; Elizabeth Tranter, MD, Principal Investigator — Hammersmith Medicines Research
Locations (3):
- United Kingdom (3):
  - Hammersmith Medicines Research, London
  - Respiratory Clinical Trials, London
  - Medicines Evaluation Unit, Manchester

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2012-001483-29